CLINICAL TRIAL: NCT02524613
Title: Prospective Bone Marrow Biopsy Safety and Efficacy Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Jacobi Medical Center (Other)
Responsible Party: Principal Investigator, Weijuan Li, MD, MS, Jacobi Medical Center
Other Study IDs: 2015-4653
Record Dates: First submitted 2015-08-06; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Bone Marrow

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Pelvis CT scan

SUMMARY:
Bone marrow biopsy is a frequently performed procedure to diagnose and evaluate hematologic diseases. It is estimated that over 700,000 bone marrow procedures (BMP's) are performed annually in the U.S. Most of them are performed by practicing hematologists/oncologists in their offices or hospitals. However, a significant number are performed by hematologists-in-training (H-I-T's) in teaching hospitals. However, the incidences of complications associated with bone marrow biopsy are largely unknown. This study has two goals:

1. The first goal is to objectively determine by CT and clinical assessment, the actual risk to patients of the bone marrow biopsy and the rate of pelvic injury in an unselected group of hematology patients requiring a bone marrow biopsy, as performed by hematologist-in-training.
2. The second goal is to determine the quality of bone marrow biopsies obtained, using the lateral angulation technique.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a hematological or oncological condition which requires a bone marrow aspiration and biopsy procedure, and no alternative procedures are available for diagnosis, staging, monitoring or follow up of their disease.
2. Subjects must be able to understand the risks/benefits and provide written informed consent to participate in the study, and be willing to participate in all required study activities for the duration of the study.
3. Subjects must be 40 years of age or older.

Exclusion Criteria:

1. Patients unable to give consent because they are decisionally impaired or have a language barrier that cannot be overcome.
2. Psychiatric or cognitive illness or recreational drug/alcohol abuse that, in the opinion of the investigator would effect subject safety and/or compliance.
3. Patients with uncontrolled bleeding disorders.
4. Pregnant and lactating females (due to radiation exposure during the CT scans).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult hematology patients who have just completed an elective bone marrow biopsy will be considered eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Complication rates associated with bone marrow biopsy | 5 days after the bone marrow biopsy
  Complications will be assessed by a modified pelvic CT
Quality of bone marrow biopsy | 5 days after the bone marrow biopsy
  Length of the bone marrow biospy specimen in mm is measured by a pathologist blindly

REFERENCES:
- [Derived] Reed LJ, Attarian S, Olson TR, Singh S, Shestopalov A, Friedman EW. Feasibility and safety of targeting the anterior superior iliac spine to perform a bone marrow procedure: a prospective, clinical study. J Clin Pathol. 2018 Dec;71(12):1116-1119. doi: 10.1136/jclinpath-2018-205309. Epub 2018 Oct 23. PMID 30352912
- [Derived] Attarian S, Reed L, Singh S, Shestopalov A, Singh AP, Budhathoki A, Abi-Aad S, Shah UA, Kim S, Bachiashvili K, Elrafei T, Li W, Yee C, Friedman EW. Visualization of the bone marrow biopsy needle track. Am J Hematol. 2018 Mar;93(3):E60-E61. doi: 10.1002/ajh.24985. Epub 2017 Dec 6. No abstract available. PMID 29168229
- [Derived] Reed L, Attarian S, Pendurti G, Singh AP, Budhathoki A, Abi-Aad S, Shah UA, Kim S, Bachiashvili K, Moon JY, Kim M, Elrafei T, Alexis K, Strakhan M, Li W, Friedman E. Targeting the anterior superior iliac spine yields significantly longer bone marrow cores. J Clin Pathol. 2018 Feb;71(2):172-173. doi: 10.1136/jclinpath-2017-204686. Epub 2017 Aug 26. PMID 28844037